CLINICAL TRIAL: NCT04817319
Title: Risk of Contamination by COVID-19 During Oral Care With Aerosolization
Acronym: Bu-Covid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP200933
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Contamination by COVID 19 During Oral Care
Keywords: COVID-19; Dental care; Aerosols
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Major patients diagnosed with Covid + requiring oral care. (Experimental)
  Interventions: Procedure: Oral care with/without aerosolization

INTERVENTIONS:
Procedure: Oral care with/without aerosolization — These treatments involve instruments that produce aerosolization: ultrasonic scaler, rotary instrumentation for caries care, dental extraction, tooth polishing.
  These care correspond to examinations of the oral cavity, intraoral X-rays or even periodontal pocket probing.

SUMMARY:
The sudden Covid-19 pandemic has led all healthcare workers to adapt to an unprecedented situation by continuing to provide care while protecting themselves and their patients. Medical care with aerosolization systems is particularly of risk because of the strong propagation of the droplets they generate, especially during oral care. Considering the high risk of transmission of the SARS-CoV-2 virus in dental structures remain essential and still very challenging. The need to put in place care procedures to protect the nursing staff and patients is definitely more than necessary. Dental protection equipments against this emergent virus have progressively integrated daily practice, but, to the knowledge of the investigators, no study has precisely evaluated their efficiency.

The main objective of this study is to estimate the risk of dental practitioners to be contaminated by SARS-CoV-2 during dental procedures with or without aerosolization procedures.

For this, after their informed consent, vaccinated dental practitioners or practitioners with a positive covid serological tests of the dental department of Charles Foix hospital will receive individually forty to fifty COVID+ patients. COVID + patients will be included a maximum of one week after the diagnosis of the pathology. Patient care will be determined and performed according to standard practice as part of their standard management and without interference with the study. The usual measures to protect caregivers. The included patients will undergo an oral dental procedure either with aerosolisation or not. Then, SARS-CoV 2 samples will be collected using viral swabs on different spots, followed by detection and quantification by PCR. Swabbing will be achieved on:

* The facial skin, nasal, ocular and oral mucosa of the practitioners.
* The protection equipment of the practitioners (FFP2 masks, visors,surgical calot,gloves) .
* The environment (dental Chair, surgical light, turbine, contra-angle, on the ground..) The presence of viral loads in areas used by COVID + patients will be evaluated by PCR after swabbing.

The study will provide insight into the risk of SARS-CoV 2 contamination for practitioners performing dental procedures in COVID + patients. This risk will be assessed at the level of the facial skin and oral mucous membranes, which are the doors of entry of the virus.

This study will thus make it possible to assess the protective capacity of the protection protocol implemented in investigators' department in this epidemic situation. This will be assessed depending on whether or not aerosolization is used, its type and the nature of the ventilation in the operating room.

DETAILED DESCRIPTION:
Introduction The outbreak of severe acute respiratory syndrome with coronavirus 2 (SARS-CoV 2) in Wuhan, China, in December 2019, quickly turned into a global pandemic (12 March 2020, WHO) leading most countries to take exceptional health measures. Indeed, in the absence of a proven treatment against COVID-19, the preventive approach aimed at reducing the risk of transmission; containment, barrier measures, has been put forward in many countries.

In this context, healthcare workers are in the front line of SARS-CoV 2 and present a high risk of contamination. Among them, dentists have been identified as the health professionals most at risk of contamination by SARS-CoV2. Indeed, SARS-CoV2 is transmitted, directly or indirectly, by respiratory secretions via airborne particles called aerosols. The virus can thus be detected in secretions from the nasopharynx but also in saliva.

For the specialities covering the ENT sphere, the main routes of contamination are blood, saliva droplets and direct contact with the patient. For SARS-CoV 2, its high contagiousness adds to the risk factors related to the proximity of the oral cavity of patients during care. Contact with nebulisers such as ultrasound (used for scaling), turbines or contra-angles (used for tooth and jawbone milling) contribute to aerosol and splash formation. Aerosols remain suspended in the air for several minutes, and can therefore increase the risk of SARS-CoV2 infection. Aerosols from an infected patient can increase the risk of infection for ENT professionals and the risk of spreading the virus to other patients.

For example, oral health care has been reduced to emergencies only in many countries. The same is true in France where the recommendations of the ARS and the Order of Dental Surgeons have followed the same objectives .

Globally, the only available studies on dental care during COVID have reviewed the organisation and procedures in place in dental departments.

However, no study has assessed the specific risk of SARS-CoV 2 contamination for practitioners, especially for procedures performed with aerosolisation.

It is therefore essential to assess the risk of contamination for practitioners performing care on a cohort of COVID+ patients.

Research hypothesis The hypothesis of this research project is that the protection protocols (patient circuit, personal protective equipment (PPE)), implemented in the oral medicine department of the Charles Foix Hospital, effectively protect oral health care workers from a Covid-19 infection, whether for care with or without nebulisation (aerosolisation). These protocols, once validated in this study, would be applicable and can be generalised.

Description of the study population and rationale for its choice The patients: COVID+ patients who will undergo a dental procedure will be included at most one week after the diagnosis of the pathology. This is because the viral load is increased in the saliva of an infected patient within this time frame (would increase the risk of infection in oral health professionals .

Practitioners: these are the dental surgeons, oral surgeons, interns and externs in dental surgery affiliated with the odontology department of the Charles Foix Hospital (APHP). These practitioners are at risk of contamination during aerosolisation procedures.

Description of procedures or products used in accordance with standard practice The patients included will all undergo an oral procedure with or without aerosolisation.

The care of COVID+ patients follows the procedure established in the Charles Foix during this health crisis. Patient care will be determined and carried out according to usual practice as part of their standard care and without interference with the study. The usual protective measures for caregivers include: FFP2 masks, visors, gloves, caps, and gowns. Hydro-alcoholic rubbing before and after care is performed systematically

The risk of contamination of practitioners will be assessed in the following way:

* A description of the projection areas (and therefore contamination) on the PPE and the environment. For this purpose, fluorescein will be added to the mouthwash for non-aerosolised procedures and to the irrigation system for aerosolised procedures.
* The procedure rooms will be exposed to a UV lamp. Pictures will be taken to visualise the contaminated areas. An estimate of the level of contamination for each procedure will be made by counting the number of fluorescent sprays per unit of total area.
* At the end of each procedure, surface swabs will be taken from the PPE (visors and gloves) as well as from the facial skin and mucous membranes (oral, ocular, nasal) of the practitioner, followed by detection and quantification by PCR (main evaluation criterion).
* The presence of viral loads on the areas used by COVID+ patients will be assessed by PCR after swabbing.

Biological collection The RNA samples taken during the research will not be the subject of a biological collection.

During the research, the collections will be kept and analysed in Cordeliers laboratory (INSERM U1138 unit) under the responsibility of François Ferré. They will be destroyed at the end of the PCR analyses.

Risks and vigilance Adverse effects observed in patients participating in the research are reported by the investigators in accordance with the local vigilance plans set up in the context of healthcare activities.

Data management The patients' medical and dental data will be collected on the same day on a dedicated database (Excel type).The PCR data of the practitioners will be collected at the Cordeliers Research Centre and stored on a dedicated database (Excel type), the PCR results will then be sent to Dr Ferré (Dispose).

A correspondence database (Excel file) linking the subject's identity to the pseudonymised identifier will be kept within the hospital department in a secure computer file on a single workstation identified and secured by the password of the coordinating investigator.

In accordance with GCP :

* the sponsor is responsible for obtaining the agreement of all parties involved in the research to ensure direct access to all research sites, source data, source documents and reports for quality control and audit purposes by the sponsor,
* the investigators will make available to the persons in charge of monitoring, quality control, in the event of an audit of the research involving the human person, the documents and individual data strictly necessary for this control, in accordance with the legislative and regulatory provisions in force Source documents, defined as any original document or object that can be used to prove the existence or accuracy of a data item or fact recorded during the research, will be kept for 15 years by the investigator or by the hospital in the case of a hospital medical file.

Within the framework of the research, additional examinations (serological examinations linked to the COVID status of patients, biological examinations, imaging, etc.) will be scanned and kept in the ORBIS computerised medical file dedicated to the patient.

The persons responsible for the quality control of research involving the human person (article L.1121-3 of the public health code), will take all the necessary precautions to ensure the confidentiality of the information relating to the research, to the persons who take part in it and in particular with regard to their identity as well as the results obtained.

These persons, in the same way as the investigators themselves, are subject to professional secrecy (in accordance with the conditions defined by articles 226-13 and 226-14 of the penal code).

During research involving the human person and at its conclusion, the data collected on the persons involved and transmitted to the sponsor by the investigators (or any other specialist) must be made non-identifying.

Under no circumstances should the names of the persons concerned or their addresses appear in clear text. Only the coded (pseudonymised) identifiers of the subjects included will be recorded.

The sponsor will ensure that each person who takes part in the research has given his/her consent to access his/her individual data which are strictly necessary for the quality control of the research.

The AP-HP is the owner of the data and no use or transmission to a third party can be made without its prior agreement.

Statistical aspects Seventy odontological procedures will be evaluated in the study. This number of 70 procedures was set to allow a sufficiently informative estimate of the proportions of procedures resulting in muco-cutaneous contamination of the practitioners who performed the procedures. Thus, if the observed frequency is 10% (7 out of 70), the estimate of the percentage will be known with a precision close to 10% IC95% = [4%; 19.5%], and under the expected hypothesis that no contamination would be observed among 70 procedures, the 95% confidence interval will then make it possible to exclude a risk of contamination higher than 5% (IC95%=[0%; 5. 1%]) and thus to be able to conclude with robustness that there is a very low risk of contamination of odontological procedures in COVID+ patients under the usual protective conditions.

Statistical analyses will be performed at the end of the inclusion period (6 months). The URC of the Pitié-Salpétrière Hospital will be responsible for the statistical analysis of the data from the study.

Description of the statistical methods

* Subgroup analyses by Cochran test:
* Ocular mucosa/Nasal mucosa/Oral mucosa/Facial skin
* Face / PPE
* Oral procedures with aerosolization/ Oral procedures without aerosolization
* Ventilated rooms/ Non-ventilated rooms

Ethical and legal aspects The Assistance Publique - Hôpitaux de Paris is the promoter of this research and by delegation the Clinical Research and Innovation Department (DRCI) is responsible for its missions, in accordance with article L.1121-1 of the public health code. Assistance Publique - Hôpitaux de Paris reserves the right to interrupt the research at any time for administrative reasons.

The practitioner and the patient who meet the selection criteria can only be included in the study after they have received the study information notes and have indicated that they do not object to participating.

In accordance with article L1121-1-1 of the Public Health Code, no non-interventional research may be performed on a person if he or she has objected to it after having been given the information provided for in article L11222-1 of the same code.

A copy of the information document is given to the person prior to participation in the research.

The information given to the subject will be notified in his or her medical file.

The investigator or the qualified person who collects the subject's non-opposition will record it in his/her medical file.

Requesting an opinion from the Committee for the Protection of Persons (CPP) The AP-HP, as the promoter, obtains a favourable opinion from the relevant CPP for research that meets the definition of 3° of article L.1121-1 of the Public Health Code, prior to its implementation, within the framework of its competences and in accordance with the legislative and regulatory provisions in force.

FUNDING A financial contribution from the Fondation des Gueules Cassées is expected to finance the purchase of reagents necessary for the PCR.

ELIGIBILITY:
Inclusion Criteria:

COVID + patients

* Over the age of 18
* Tested positively a maximum of one week before inclusion
* Requiring oral care
* Affiliates or beneficiaries of Social Security • Informed and not opposed to participating in the research

Practitioners

* Age under 65
* Absence of comorbidity (hypertension, obesity, diabetes)
* Informed and not opposed to participating in the research

Exclusion Criteria:

COVID + patients

* State of health incompatible with oral care.
* Patient under guardianship / curators
* Pregnant or breastfeeding patients
* Pregnant / breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the risk of skin and mucous membrane contamination of practitioners during oral care performed on patients diagnosed with COVID +. | 6 months after the beginning of the study
  Percentage of odontological procedures leading to the detection of SARS-CoV 2 on the face (skin surface and facial mucous membranes) of practitioners performing procedures on COVID + patients

SECONDARY OUTCOMES:
Determine the presence of SARS-CoV 2 on the face and facial mucous membranes of practitioners after the dental procedure depending on whether: • the procedure involves aerosolization (turbine, ultrasonic scaler,…), | 6 months after the beginning of the study
  Calculation of the percentages of procedures leading to the detection of SARS-CoV 2 on the face (skin surface and facial mucous membranes) of the practitioners performing the interventions depending on whether the procedure involves aerosolization or not.
Determine the presence of SARS-CoV 2 on the face and facial mucous membranes of practitioners after the dental procedure depending on whether: • the procedure does not involve aerosolization (intraoral examination, intraoral X-ray, biopsy) | 6 months after the beginning of the study
  Calculation of the percentages of procedures leading to the detection of SARS-CoV 2 on the face (skin surface and facial mucous membranes) of the practitioners performing the interventions depending on whether the procedure involves aerosolization or not.
Determine the presence of SARS-CoV 2 on personal protective equipment (PPE) depending on whether: • the procedure involves aerosolization (contra-angle, ultrasonic scaler), | 6 months after the beginning of the study
  Calculation of the percentages of procedures leading to the presence of SARS-CoV 2 detected on PPE depending on whether the procedure involves aerosolization or not
Evaluate the risk of contamination of practitioners, PPE and surfaces depending on the type of aerosolization used (contra-angle, ultrasonic scaler) | 6 months after the beginning of the study
  Comparison of viral loads and projections on PPE and the face (skin surface and facial mucous membranes) according to the aerosolizations used (contra-angle, ultrasound)
Evaluate the risk of contamination of practitioners, PPE and surfaces depending on the type of aerosolization used (contra-angle, ultrasonic scaler) | 6 months after the beginning of the study
  Comparison of the exposure time.
Evaluate the presence of viral loads in areas used by COVID + patients | 6 months after the beginning of the study
  PCR test on the surfaces of areas used by COVID + patients

CONTACTS AND LOCATIONS:
Locations (1):
- service d'odontologie, Hôpital Charles Foix, Ivry-sur-Seine, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.